CLINICAL TRIAL: NCT02660723
Title: To Investigate the Impact of Aging on Cytokine and Chemokine Production by Peripheral Blood Immune Cells
Brief Title: Impact of Aging on Cytokine Production by Innate Immune Cells
Acronym: Cytokinage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-PP-07
Record Dates: First submitted 2015-11-30; First posted 2016-01-21 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-02

CONDITIONS: Healthy
Keywords: M01.774.500; Volunteers
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy Volunteers (Other): A catheter will be introduced in the arm vein and 14 ml of blood will be drawn in one 4 ml dry tube, one 5 ml heparinized tube for cell count and 5 1 ml TruCulture tubes.
  Interventions: Other: Healthy Volunteers

INTERVENTIONS:
Other: Healthy Volunteers — A catheter will be introduced in the arm vein and 14 ml of blood will be drawn in one 4 ml dry tube, one 5 ml heparinized tube for cell count and 5 1 ml TruCulture tubes.
  Other Names: blood test

SUMMARY:
The main goal of this study is to investigate the impact of aging on the responsiveness of peripheral blood immune cells. To this aim, the investigators will take advantage of a recently described syringe-based assay system that can reproducibly assess induced, innate or adaptive immune responses. Briefly, a total of 50 healthy volunteers will participate to this study: 25 will be older than 18 and younger than 30, and 25 will be older than 55. A total of 14 ml of blood will be drawn including 5 X 1 ml in TruCulture™ tubes containing poly(I:C), R-848, LPS, CpG, or no stimulus, respectively. After 22 hours of incubation at 37°C, cellular supernatants will assessed for levels of 10 different chemokines using a MesoScaleDiscovery multiplexing platform.

ELIGIBILITY:
Inclusion Criteria:

* volunteers will be invited to settle an appointment with the Nice University Hospital (CHU de Nice) Research Clinical Center (CRC).
* being between 18 and 30 year-old (group Y) or being older than 55 year-old (group O),
* ability to understand and speak French,
* being registered at the Social Security,
* acceptance to be serologically tested for HIV and HVC,
* considered healthy based on both past medical records and the clinical examination performed at the inclusion visit,
* exhibiting a body mass index (body mass divided by the square of their height) comprised between 18.5 and 30.0 kg/m2.

Exclusion Criteria:

* having participated to a drug clinical trial since less than 3 months,
* having traveled to a tropical or a sub-tropical country over the past 3 months,
* being pregnant or a lactating mother (for women),
* having performed intensive physical exercise over the past 12 hours,
* following a specific diet for medical reasons,
* over-drinking, i.e. more that 50 g of pure alcohol every day,
* having taken an immuno-suppressive or immuno-modulatory drug over the past two weeks, or for at least 14 consecutive days over the past 6 months,
* having been vaccinated over the past 3 months,
* declaring not being on an empty stomach for less than 12 hours,
* having received a blood transfusion or intravenous immunoglobulins over the past 3 months,
* declaring being HIV- or HVC- positive,
* having suffered from an infection since less than 3 weeks,
* exhibiting a positive urine pregnancy test at the inclusion visit,
* suffering from a severe/chronic/relapsing pathology, i.e. inflammatory bowel disease, psoriasis, atopic dermatitis, rheumatoid arthritis, multiple sclerosis, type I or type II diabetes, Parkinson's disease, and (p) having been diagnosed with a cancer and not being in a remitting period for less than 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
CCL2 levels | at first day
  Compare CCL2 levels in the supernatants of poly(I :C)-stimulated whole blood cells between volunteers aged from 18 to 30 years and volunteers older than 55

SECONDARY OUTCOMES:
Other CCL levels | at first day
  Compare CXCL8 (IL-8) levels in the supernatants of poly(I :C)-stimulated whole blood cells between volunteers aged from 18 to 30 years and volunteers older than 55

CONTACTS AND LOCATIONS:
Overall Officials: Passeron Thierry, PhD, Principal Investigator — CHU de Nice, Service de Dermatologie
Locations (1):
- CHU de Nice, CRC, Hôpital de l'Archet 151 route de saint-antoine de ginestière, Nice, Alpes-Maritimes, France

IPD SHARING:
Plan to Share IPD: No